CLINICAL TRIAL: NCT02551588
Title: Calcified Aortic Valve Stenosis (AVS). Markers of Fibrosis Using Cardiac Magnetic Resonance
Brief Title: Valvular Aortic Stenosis: Study of Myocardiac Fibrosis by Magnetic Resonance Imagery
Acronym: RACINE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081112
Record Dates: First submitted 2015-09-04; First posted 2015-09-16 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Aortic Valve Stenosis
Keywords: fibrosis; Magnetic resonance imaging
MeSH Terms: conditions — Aortic Valve Stenosis; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Valvular aortic stenosis surgery: Patients with symptomatic AVS had indication for surgery. They were proposed to have per procedure cardiac biopsy.
  They were followed when possible one year after surgery.
  Interventions: Procedure: Valvular aortic stenosis surgery
- Valvular aortic stenosis without surgery: These patients with asymptomatic AVS had no indication for surgery. They were followed when possible one year after inclusion.
- Control subject: Patients without history of cardiac infarction, primary or secondary myocardiopathy or of radiotherapy or chemotherapy.

INTERVENTIONS:
Procedure: Valvular aortic stenosis surgery — Dilatation of Valvular aortic stenosis
  Groups: Valvular aortic stenosis surgery

SUMMARY:
Aortic valve stenosis (AVS) is the most frequent valvular disease. The severity of the obstruction of the left ventricle (LV) is essentially analyzed today by echocardiography Doppler, which assesses two key markers that are aortic valve pressure gradient and the aortic valve area. however these marker are a poor reflect of the clinical severity of AVS. The aim of the study is to validate new markers assessing cardiac fibrosis that might best or complementary markers.

DETAILED DESCRIPTION:
To validate new markers assessing cardiac fibrosis three groups of subjects were studied in controls subjects and patients with AVS in order to :

1. Analyze myocardial fibrosis markers in MRI, the degree of hypertrophy, remodeling and wall shear stress in a control population and in three groups of subjects to RA progressively increasing risk: asymptomatic subjects without symptomatic subjects LV dysfunction, symptomatic patients with LV dysfunction. The factors favoring the appearance of fibrosis observed in MRI will be analyzed on all subjects.
2. To validate these fibrosis markers estimated by MRI by histological analysis of biopsies performed in patients undergoing aortic valve replacement.
3. Monitoring compliance with the distribution of markers of fibrosis and wall stress estimated on Initial MRI are factors of aggravation or not improved function and / or remodeling remote myocardial. Public hospitals in Paris

ELIGIBILITY:
PATIENTS :

Inclusion Criteria:

* Echocardiography considered as normal and / or age-related
* Patients who have received prior clinical examination
* Patient receiving a social security scheme or entitled, or CMU
* After having giving written informed consent.
* Patients symptomatic with indication of surgery (group surgery) or not

Exclusion Criteria:

* With one of the following cardiac abnormalities: atrial fibrillation, more than moderate either aortic or mitral valve regurgitation
* Heart valve surgery history (aortic, mitral, tricuspid and pulmonary).
* Indication for cardiac surgery other than on the aortic valve.
* Usual counter-indications of MRI: Pace-maker, defibrillator, metallic objects including gadolinium allergy.
* Patients with severe renal insufficiency with a clearance <30 ml / min estimated by the Cockcroft & Gault formula.
* Patient who cannot be followed over the duration of a year.

CONTROLS (healthy volunteers)

Inclusion criteria:

* Normal EKG
* Echocardiography considered normal and / or age-related
* Patients who have received prior clinical examination
* Patient receiving a french national social security
* After having obtain written informed consent.

Criteria for non-inclusion

* History of known or detectable infarction on EKG
* Known primary or secondary cardiomyopathy or detectable on echocardiography
* Thoracic radiotherapy or chemotherapy history
* Subject with usual contra-indications of MRI: claustrophobia, metallic objects.
* Patients with significant renal insufficiency with a clearance <90 ml / min estimated by the Cockcroft & Gault formula.
* Subject who could be planned for 2 CMR within two weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Valvular Aortic Stenosis with or without surgery (symptomatic patients) or controls
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
prevalence of myocardial fibrosis in MRI in patients with AVS | At one year
  Indices of myocardial fibrosis will been analysed as combined criteria to analyse myocardial fibrosis

SECONDARY OUTCOMES:
comparison of these markers with myocardial histology | At inclusion and at one year
  Fibrosis estimated by MRI will be compared to fibrosis on myocardial biopsy symptomatic patients with surgery only)
Correlation with Doppler Echocardiography Assessment, and wall stress estimate by using both cardiac MR and carotid artery pressure (applanation tonometry) | At inclusion and at one year
  Correlation of MRI with known markers of ventricular hypertrophy

CONTACTS AND LOCATIONS:
Overall Officials: Elie MOUSSEAUX, MD, PhD, Principal Investigator — Departement of Radiology, Hopital Europeen Georges Pompidou, Paris, France. Tel: +33 1 56 09 37 09. E-mail: elie.mousseaux@egp.aphp.fr
Locations (1):
- Departement of Radiology, Hopital Europeen Georges Pompidou,, Paris, France